CLINICAL TRIAL: NCT04005170
Title: A Phase II Trial of Combination of Toripalimab and Definitive Chemoradiotherapy in Esophageal Squamous Cell Carcinoma
Brief Title: Combination of Toripalimab and Chemoradiotherapy in Esophageal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mian XI (Other)
Responsible Party: Sponsor-Investigator, Mian XI, Associate professor, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TORIDEFEC
Record Dates: First submitted 2019-06-26; First posted 2019-07-02 (Actual); Last update posted 2022-08-23 (Actual); Status verified 2022-08

CONDITIONS: Unresectable Esophageal Cancer
Keywords: Esophageal squamous cell carcinoma; Definitive chemoradiotherapy; Toripalimab; Clinical complete response
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — toripalimab; TP protocol; Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PD-1 group (Experimental): All patients will receive standard fractionation radiation therapy (RT) scheme: 50.4 Gy in 28 fractions over 5-6 weeks, concurrently with 5 cycles of paclitaxel/cisplatin (paclitaxel 50mg/m2 and cisplatin 25 mg/m2) on days 1, 8, 15, 22, 29 and 2 cycles of toripalimab 240 mg on days 1, 22 followed by a maintenance phase of toripalimab IV 240 mg every 3 weeks for up to 1 year.
  Interventions: Drug: Toripalimab; Drug: Paclitaxel/Cisplatin; Radiation: Intensity-modulated radiotherapy

INTERVENTIONS:
Drug: Toripalimab — Patients received toripalimab 240 mg on days 1 and 22 during radiotherapy followed by a maintenance phase of toripalimab IV 240 mg every 3 weeks for up to 1 year.
  Other Names: JS-001
Drug: Paclitaxel/Cisplatin — Patients received 5 cycles of paclitaxel/cisplatin (paclitaxel 50mg/m2 and cisplatin 25 mg/m2) on days 1, 8, 15, 22, 29 during radiotherapy.
  Other Names: TP
Radiation: Intensity-modulated radiotherapy — All patients received external-beam radiation using intensity-modulated radiotherapy. The prescribed dose is 50.4 Gy in 28 fractions over 5-6 weeks.
  Other Names: IMRT

SUMMARY:
Definitive chemoradiotherapy (CRT) is the standard treatment option for unresectable esophageal cancer (EC). However, as high as more than 40% of EC patients experienced locoregional recurrence after concurrent CRT. Immunotherapy targeting the PD-1/PD-L1 checkpoints has demonstrated promising activity in advanced EC. The aim of this study was to evaluate the efficacy and safety of the combination of toripalimab (an anti-PD-1 antibody) combined with definitive CRT in locally advanced esophageal squamous cell carcinoma (ESCC).

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed squamous cell carcinoma of the esophagus;
2. Absence of hematogenous metastasis disease, confirmed by endoscopic ultrasound (EUS) and PET-CT scan (according to UICC TNM version 8);
3. Not suitable for surgery (either for medical reasons or patient's choice);
4. Age at diagnosis 18 to 70 years;
5. No prior cancer therapy;
6. Estimated life expectancy >6 months;
7. Eastern Cooperative Oncology Group performance status ≤ 2
8. No history of concomitant or previous malignancy;
9. The function of important organs meets the following requirements: a. white blood cell count (WBC) ≥ 4.0×109/L, absolute neutrophil count (ANC) ≥ 1.5×109/L; b. platelets ≥ 100×109/L; c. hemoglobin ≥ 9g/dL; d. serum albumin ≥ 2.8g/dL; e. total bilirubin ≤ 1.5×ULN, ALT, AST and/or AKP ≤ 2.5×ULN; f. serum creatinine ≤ 1.5×ULN or creatinine clearance rate >60 mL/min;
10. Ability to understand the study and sign informed consent.

Exclusion Criteria:

1. Patients who have been treated previously with anti-tumor therapy (including chemotherapy, radiotherapy, surgery, immunotherapy, etc.);
2. Patients with hematogenous metastasis disease at diagnosis;
3. Known or suspected allergy or hypersensitivity to monoclonal antibodies, any ingredients of Toripalimab, and the chemotherapeutic drugs paclitaxel or cisplatin;
4. Patients who have a preexisting or coexisting bleeding disorder;
5. Female patients who are pregnant or lactating;
6. Inability to provide informed consent due to psychological, familial, social and other factors;
7. Presence of CTC grade ≥ 3 peripheral neuropathy;
8. A history of malignancies other than esophageal cancer before enrollment, excluding non-melanoma skin cancer, in situ cervical cancer, or cured early prostate cancer
9. A history of diabetes for more than 10 years and poorly controlled blood glucose levels;
10. Patients who cannot tolerate chemoradiotherapy due to severe cardiac, lung, liver or kidney dysfunction, or hematopoietic disease or cachexia.
11. Active autoimmune diseases, a history of autoimmune diseases (including but not limited to these diseases or syndromes, such as colitis, hepatitis, hyperthyroidism), a history of immunodeficiency (including a positive HIV test result), or other acquired or congenital immunodeficiency diseases, a history of organ transplantation or allogeneic bone marrow transplantation;
12. A history of interstitial lung disease or non-infectious pneumonia;
13. A history of active pulmonary tuberculosis infection within 1 year or a history of active pulmonary tuberculosis infection more than 1 year ago but without formal anti-tuberculosis treatment;
14. Presence of active hepatitis B (HBV DNA ≥ 2000 IU/mL or 104 copies/mL), hepatitis C hepatitis C antibody, and HCV-RNA levels higher than the lower limit of the assay).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2019-06-25 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
clinical complete response rate | 3 months after chemoradiotherapy (plus or minus 14 days)
  Tumor response was evaluated 3 months after the completion of chemoradiotherapy based on CT or PET-CT scans, endoscopy with biopsies.

SECONDARY OUTCOMES:
2-year overall survival | From date of randomization until the date of death from any cause or the date of last follow-up, whichever came first, assessed up to 24 months
  The 2-year overall survival of the whole group
2-year progression-free survival | From date of randomization until the date of death from any cause or the date of first documented disease progression whichever came first, assessed up to 24 months
  The 2-year progression-free survival of the whole group
Duration of response | From date of first CR/PR to the date of first PD according to RECIST criteria, assessed up to 24 months
  Tumor response was evaluated every two months after chemoradiotherapy according to RECIST criteria
Incidence of treatment-related adverse events as assessed by CTCAE v4.0 | From the start of treatment to 2 year after the completion of treatment
  Toxicity of treatment was evaluated according to CTCAE 4.0

OTHER OUTCOMES:
The impact of PD-L1 expression on clinical response | Baseline biopsies of primary tumor in esophagus
  To investigate the impact of programmed cell death-ligand 1 (PD-L1) expression on clinical response
The impact of IDO1 expression on clinical response | Baseline biopsies of primary tumor in esophagus
  To investigate the impact of indoleamine 2,3-dioxygenase 1 (IDO1) expression on clinical response

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guanzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fu J, Wang F, Dong LH, Zhang J, Deng CL, Wang XL, Xie XY, Zhang J, Deng RX, Zhang LB, Wu H, Feng H, Chen B, Song HF. Preclinical evaluation of the efficacy, pharmacokinetics and immunogenicity of JS-001, a programmed cell death protein-1 (PD-1) monoclonal antibody. Acta Pharmacol Sin. 2017 May;38(5):710-718. doi: 10.1038/aps.2016.161. Epub 2017 Mar 20. PMID 28317872
- [Background] Tang B, Yan X, Sheng X, Si L, Cui C, Kong Y, Mao L, Lian B, Bai X, Wang X, Li S, Zhou L, Yu J, Dai J, Wang K, Hu J, Dong L, Song H, Wu H, Feng H, Yao S, Chi Z, Guo J. Safety and clinical activity with an anti-PD-1 antibody JS001 in advanced melanoma or urologic cancer patients. J Hematol Oncol. 2019 Jan 14;12(1):7. doi: 10.1186/s13045-018-0693-2. PMID 30642373
- [Background] Zhou S, Zhao L, Liang Z, Liu S, Li Y, Liu S, Yang H, Liu M, Xi M. Indoleamine 2,3-dioxygenase 1 and Programmed Cell Death-ligand 1 Co-expression Predicts Poor Pathologic Response and Recurrence in Esophageal Squamous Cell Carcinoma after Neoadjuvant Chemoradiotherapy. Cancers (Basel). 2019 Feb 1;11(2):169. doi: 10.3390/cancers11020169. PMID 30717285
- [Derived] Wang R, Ling Y, Chen B, Zhu Y, Hu Y, Liu M, Yang Y, Zhang L, Lv Y, Liu S, Li Q, Xi M. Long-term survival and post-hoc analysis of toripalimab plus definitive chemoradiotherapy for oesophageal squamous cell carcinoma: insights from the EC-CRT-001 phase II trial. EClinicalMedicine. 2024 Aug 30;75:102806. doi: 10.1016/j.eclinm.2024.102806. eCollection 2024 Sep. PMID 39281099
- [Derived] Zhu Y, Wen J, Li Q, Chen B, Zhao L, Liu S, Yang Y, Wang S, Lv Y, Li J, Zhang L, Hu Y, Liu M, Xi M. Toripalimab combined with definitive chemoradiotherapy in locally advanced oesophageal squamous cell carcinoma (EC-CRT-001): a single-arm, phase 2 trial. Lancet Oncol. 2023 Apr;24(4):371-382. doi: 10.1016/S1470-2045(23)00060-8. PMID 36990609